CLINICAL TRIAL: NCT02313714
Title: Effects of Neuromuscular Electrical Stimulation in Patients With Congestive Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Orlando Petrucci, MD, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ENESPHF
Record Dates: First submitted 2013-11-27; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Heart Failure
Keywords: heart failure, heart transplant, electrical stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular stimulation (Experimental): The patients will receive electric muscular stimulation with a Russian current protocol twice a week for 7 weeks.
  Interventions: Device: stimulation wave (2.5 kHz, burst at 50Hz, on/off: 3/9 sec),
- Sham Group (Placebo Comparator): The patients will receive very low electric muscular stimulation with a no biological or clinical effects
  Interventions: Device: Sham

INTERVENTIONS:
Device: stimulation wave (2.5 kHz, burst at 50Hz, on/off: 3/9 sec), — All patients in the treatment arm will receive electric muscular stimulation with a Russian current protocol twice a week for 7 weeks.
  Other Names: Neuromuscular stimulation
  Arms: Neuromuscular stimulation
Device: Sham — very low electric muscular stimulation
  Arms: Sham Group

SUMMARY:
This study intends to treat patient with congestive heart failure that are maximized their pharmacological treatment and at heart transplant wait list.

All patients in the treatment arm will receive electric muscular stimulation with a Russian current protocol twice a week for 7 weeks.

The outcome will be assessed by the improvement in quality of life and functional capacity.

DETAILED DESCRIPTION:
The neuromuscular electrical stimulation (NMES) has been used as adjuvant treatment in patients with end-stage congestive heart failure. Those patients are limited to perform conventional physical activity and adherence to any every day protocols frequency. The aim of this study was evaluated the effect on functional status and quality of life after NMES treatment using Russian stimulation wave solely twice a week during five weeks period in patients waiting for a heart transplant.

Inclusion criteria:

Age between 30 to 80 years old Congestive heart failure in NYHA class III or IV Ejection fraction lower than 35% Stable clinical status Full pharmacologic treatment

Exclusion criteria:

Unstable angina Ventricular arrhythmia intermittent lameness Inferior limb amputation

Protocol Design:

Patients at waiting list for heart transplant will be invited to participate on protocol of NMES using Russian stimulation wave (2.5 kHz, burst at 50Hz, on/off: 3/9 sec), named NMES group or sham stimulation, named control group. The NMES will be applied for 50 minutes, twice a week on both quadriceps femoral muscles during 7 weeks. The patients will be evaluated every week for distance walked during six minutes walk test (6MWT), heart rate variability, and functional status according to New York Heart Association. All patients were evaluated at the beginning and after completion of the protocol for quality of life with Minnesota Living with Heart Failure Questionnaire (LHFQ).

ELIGIBILITY:
Inclusion Criteria:

* patients on waiting list for heart transplant

Exclusion Criteria:

* patients that won't accept to participate in the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Improvement on distance walked in the six minute walk test | after 7 weeks of first inttervention

SECONDARY OUTCOMES:
Improvement on quality of life | 7 weeks after first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carolina Sacilotto, MsC, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil